CLINICAL TRIAL: NCT07180303
Title: A Community-Based Cluster Randomized Trial Evaluating a Colorectal Cancer Screening Program Integrated Within the Rural Primary Healthcare System in China
Brief Title: Colorectal Cancer Screening in Chinese Rural Communities
Acronym: CRC-RPHC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: RuralCRC Screen
Record Dates: First submitted 2025-08-31; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer
Keywords: Screen; Integrated CRC Screening Program
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated CRC Screening Program (Experimental): * Provide remote training courses covering the latest colorectal cancer screening guidelines, methods for identifying high-risk individuals and their standards of care, as well as dietary intervention strategies.
  * Offer ongoing support services, such as regular knowledge updates and technical consultations.
  Interventions: Other: Remote training courses covering the latest CRC screening guidelines, identification of high-risk individuals and their standard of care, and dietary intervention strategies. Ongoing support services,
- Standard Care / Usual Practice (Sham Comparator): Current opportunistic screening practices within the rural primary healthcare system.
  Interventions: Other: Continuation of routine healthcare services without any additional training interventions.

INTERVENTIONS:
Other: Remote training courses covering the latest CRC screening guidelines, identification of high-risk individuals and their standard of care, and dietary intervention strategies. Ongoing support services, — Remote training courses covering the latest CRC screening guidelines, identification of high-risk individuals and their standard of care, and dietary intervention strategies.
  Ongoing support services, such as regular knowledge updates and technical consultations.
  Arms: Integrated CRC Screening Program
Other: Continuation of routine healthcare services without any additional training interventions. — Continuation of routine healthcare services without any additional training interventions.
  Arms: Standard Care / Usual Practice

SUMMARY:
Colorectal cancer (CRC) is one of the most common malignant neoplasms significantly impacting population health and longevity. With the transformation of lifestyle and dietary patterns among Chinese residents, coupled with an increasingly aging population, both the incidence and mortality rates of CRC in China have exhibited a sustained upward trend. CRC often presents with insidious onset; the five-year survival rate for patients diagnosed at intermediate or advanced stages remains below 15%. In contrast, early diagnosis and treatment can achieve a five-year survival rate exceeding 90%. Furthermore, population-based CRC screening in mainland China is still in its nascent stages. Although preliminary, small-to-medium-scale screening programs have been implemented in certain regions, participation rates in risk assessment questionnaires and fecal occult blood testing remain suboptimal, attributable to regional disparities and variations in cultural and educational backgrounds. Moreover, adherence to the pivotal diagnostic procedure-colonoscopy-within screening programs is notably low, estimated at approximately 20% to 30%. Consequently, more refined and scientifically grounded mobilization and educational campaigns are critically important to enhance participation in population-based CRC screening initiatives.

DETAILED DESCRIPTION:
**1. Background and Objectives** This study aims to investigate, through a cluster randomized controlled trial (RCT), whether remote training for primary care physicians can effectively enhance the accessibility and adherence to colorectal cancer (CRC) screening. Specifically, the intervention group will receive professional training on CRC screening guidelines, standards of care for high-risk individuals, and dietary interventions, while the control group will receive no additional training. The ultimate goal is to improve community residents' awareness of colorectal cancer, increase screening participation, and reduce both incidence and mortality rates.

**2. Study Design**

* **Target Population:** Fifteen natural villages within a county or city will be selected as study sites, encompassing permanent residents aged between 40 and 74 years.
* **Randomization:** A cluster randomization method will be employed to randomly assign the 15 villages to either Group A (intervention group) or Group B (control group). Each group will include at least seven villages to ensure adequate sample size.
* **Sample Size Calculation:** The required sample size will be determined based on estimated changes in screening adherence rates and other relevant parameters.

**3. Intervention**

* **Intervention Group (Group A):**
* Remote training courses covering the latest CRC screening guidelines, identification of high-risk individuals and their standard of care, and dietary intervention strategies.
* Ongoing support services, such as regular knowledge updates and technical consultations.
* **Control Group (Group B):**
* Continuation of routine healthcare services without any additional training interventions.

**4. Data Collection and Analysis**

* **Primary Outcome Measures:**
* Phase I: Improvement in colonoscopy adherence.
* Phase II: Trends in colorectal cancer incidence.
* Phase III: Long-term impact on colorectal cancer mortality.
* **Secondary Outcome Measures:** Participants' understanding of CRC prevention and control, changes in lifestyle behaviors, etc.
* **Data Analysis:** Appropriate statistical software will be used to analyze the data, comparing differences between the two groups while accounting for potential confounding factors.

**5. Potential Supplementary Aspects**

* **Community Education:** Strengthen health education activities at the community level to enhance public awareness of colorectal cancer and self-protection.
* **Cost-Effectiveness Analysis:** Conduct a cost-effectiveness analysis to evaluate the economic benefits of the intervention.
* **Ethical Considerations:** Ensure all participants are fully informed about the study's purpose and provide consent, while safeguarding individual privacy.

**6. Feasibility Assessment**

* **Resource Availability:** Confirm sufficient funding to support project operations, including development of training materials and maintenance of the technological platform.
* **Technical Readiness:** Ensure the technical requirements for remote training are met, such as stable internet connectivity and a user-friendly learning management system.
* **Personnel Training:** Ensure participating healthcare providers possess the necessary foundational knowledge and can effectively apply the acquired knowledge in clinical practice.

ELIGIBILITY:
Inclusion Criteria

1. Between 45 and 70 years old (inclusive).
2. Permanent resident within the geographic area covered by the screening program (typically defined as residing in the area for a minimum period, e.g., 6 months or more), and possessing local household registration (hukou) or residency documentation.
3. Self-reported absence of symptoms suggestive of colorectal cancer (e.g., rectal bleeding, change in bowel habits, abdominal pain, palpable abdominal mass, unexplained anemia, or unintentional weight loss).
4. No prior diagnosis of colorectal cancer or precancerous lesions (e.g., high-grade intraepithelial neoplasia, serrated lesions with dysplasia).
5. Not currently participating in another colorectal cancer-related clinical study that might interfere with the screening outcomes.
6. Willing and able to provide written informed consent, agreeing to participate in the screening program and comply with subsequent follow-up procedures (e.g., fecal testing, colonoscopy).

Exclusion Criteria

1. Previous diagnosis of colorectal cancer, history of resection of colorectal polyps (especially high-grade lesions or serrated lesions with dysplasia), or diagnosis of inflammatory bowel disease (ulcerative colitis, Crohn's disease).
2. Completion of a high-quality colonoscopy within a specified timeframe (e.g., within the past 1 year) with normal results (no polyps or only 1-2 tubular adenomas <10mm), or completion of a high-quality sigmoidoscopy within a specified timeframe (e.g., within the past 3 years) with normal results.
3. Presence of severe comorbid conditions (e.g., severe cardiac, pulmonary, hepatic, or renal insufficiency) resulting in a life expectancy of less than 10 years, or physical condition unable to tolerate colonoscopy and bowel preparation.
4. Conditions such as severe coagulopathy, recent acute myocardial infarction or stroke (e.g., within the past 3 months), or severe psychiatric illness preventing cooperation.
5. Generally excluded due to safety considerations regarding screening colonoscopy during these periods.
6. Inability to understand the study content and provide informed consent due to cognitive impairment, language barriers, or other reasons.
7. Judged by the investigator to have a very high likelihood of being lost to follow-up during the study period, making completion of the screening pathway unlikely.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in colonoscopy adherence | 1 year
  Proportion of patients undergoing colonoscopy, The proportion of patients who, after questionnaire screening and fecal occult blood testing, are indicated for colonoscopy and ultimately undergo the procedure.

SECONDARY OUTCOMES:
Trends in colorectal cancer incidence | 1 year
  Trends in colorectal cancer incidence
Long-term impact on colorectal cancer mortality | 5 year
  Long-term impact on colorectal cancer mortality (5 year OS)

CONTACTS AND LOCATIONS:
Locations (1):
- Liyang Municipal Health Commission, Liyang, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
We will provide de-identified information of all individuals included in the screening in a public database, which will be accessible through an online platform. Access will be granted upon submission of a reasonable request to the lead investigator of this study.
Supporting Information: Study Protocol, SAP
Time Frame: 2 years
Access Criteria: Access will be granted upon submission of a reasonable request to the lead investigator of this study.
URL: https://www.jiandaoyun.com/index/sem/?utm_src=ppbysem_kw42357&msclkid=1295140a61f919e5961e7cc801db36e2